CLINICAL TRIAL: NCT02103075
Title: Neuromuscular Electrical Stimulation on Median Nerve Facilitates Low Motor Cortex Excitability in Human With Spinocerebellar Ataxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Professor, Chang Gung University
Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 91-221
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-03

CONDITIONS: Spinocerebellar Ataxia
Keywords: spinocerebellar ataxia (SCA); motor evoked potential (MEP); Neuromuscular electrical stimulation (NMES); silent period; cerebellum
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- The SCA (Experimental)
  Interventions: Device: Neuromuscular electrical stimulation
- The age-matched control (Experimental)
  Interventions: Device: Neuromuscular electrical stimulation
- The young control (Experimental)
  Interventions: Device: Neuromuscular electrical stimulation

INTERVENTIONS:
Device: Neuromuscular electrical stimulation — All groups received an accumulated 30-minute NMES (25 Hz, on/off: 800ms/800ms) intervention on median nerve.

SUMMARY:
Spinocerebellar ataxia (SCA) is a hereditary disorder with movement incoordination. The ataxia performed low intra-cortical facilitation mainly due to the degenerative cerebellum. Noninvasive sensory stimulations such as peripheral electrical stimulation were reported to modulate the excitability of the motor excitability. Neuromuscular electrical stimulation (NMES) was proposed as a neuromodulation tool for the aberrant motor excitability on the SCA. This study aims to investigate the effect of NMES on the motor excitability in the SCA, and the differentiation on the central or peripheral motor excitability changed by the NMES.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Spinocerebellar ataxia
* No history of epilepsy
* No other neuromuscular disorder
* No fracture within the last six months and restricted movement on the upper extremity
* Limited trembling hand allowed for the EMG recording.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2002-08; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Central Motor Excitability | Baseline, in experiment, 0 minute, 10 minutes, and 20 minutes.
  Measure of changes in Central Motor Excitability by motor evoked potential and silent period that are measured by transcranial magnetic stimulation.
Peripheral Motor Excitability | Baseline, in experiment, 0 minute, 10 minutes, and 20 minutes.
  Measure of changes in peripheral motor excitability by Maximum M wave and H reflex

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Chen CC, Chuang YF, Yang HC, Hsu MJ, Huang YZ, Chang YJ. Neuromuscular electrical stimulation of the median nerve facilitates low motor cortex excitability in patients with spinocerebellar ataxia. J Electromyogr Kinesiol. 2015 Feb;25(1):143-50. doi: 10.1016/j.jelekin.2014.10.009. Epub 2014 Nov 1. PMID 25434572